CLINICAL TRIAL: NCT03116334
Title: Shared Genetic Influences Between Cognitive Function and Body Mass Index (BMI) in the Texas Twin Project
Brief Title: Genetic Influences Between Cognitive Function and BMI
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Alexis Wood, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-37801
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Obesity
Keywords: Obesity; BMI; executive functioning; general cognitive ability; twin study; heritability; cognition; GCTA
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the investigators will interrogate an existing data set to examine whether genetic variants contribute to an inverse association between weight status and cognitive function. Investigators hypothesize that body mass index (BMI) will be inversely related to a number of variables measuring cognitive function, and that that this inverse relation will be at least partially attributable to genetic variants which influence both BMI and cognition.

DETAILED DESCRIPTION:
Investigators will use existing data collected as part of the Texas Twin Project (TTP). TTP collected neuropsychological task data on cognition (executive functioning and general cognitive abilities) from a computerized test battery, as well as BMI data, on a sample of 869 twins. Investigators will use information from the known extent of genetic and environmental sharing between members of MZ (monozygotic; identical) and DZ (dizygotic; fraternal) twin pairs to quantify the genetic correlation between measures of cognition and BMI using biometric genetic modeling under the assumptions of the classical twin model. The specific aims are:

* To examine the association between BMI and executive functioning (EF) in a sample of 869 twin children, ages 7 to 15 years old, who participated in the Texas Twin Project (TTP)
* To gauge the specificity of EF-BMI relations relative to academic achievement and general cognitive abilities.
* To examine the relative contribution of genetic and environment influences to the inverse association between BMI and EF

ELIGIBILITY:
Inclusion Criteria:

All participants in the TTP database with executive functioning and BMI data, without a parent-reported medical disorder affecting growth

Exclusion Criteria:

Parent-reported medical disorder affecting growth More than one sibling in the dataset (if triplets are present, only two randomly selecting siblings will be included).

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Individuals from the Texas twin Project dataset, who were twins and higher-order multiples previously recruited from the Houston and Austin Metropolitan areas, via flyers, the internet (study website) and contact through public school rosters
Sampling Method: Non-Probability Sample
Enrollment: 869 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Executive functioning | 2 hours
  This measure will be derived from a computerized test battery incorporating the Animal Stroop, Stop Signal, Mickey (an anti- Trail Making, Local-Global, Plus-Minus, Digit Span Backward, Symmetry Span, Listening Recall, 2-Back, Keeping Track, and Running Memory for Letters tasks. A latent factor of variance common to all these tasks will be used to indicate "higher order executive functioning".
Body mass index | 10 minutes
  Heights and weights were measured by trained study personnel and BMI will be calculated as weight in kilograms (kg) divided by height in centimeters (cm) squared.

SECONDARY OUTCOMES:
General Cognitive Ability | 1 hour
  This was assessed using the WASI-II
Academic Achievement | 30 minutes
  This was assessed using the Woodcock-Johnson-III Calculations and Passage Comprehension tests

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This protocol involves secondary data analysis of existing studies. Data will not be shared with other investigators since they should obtain data from the primary sources.